CLINICAL TRIAL: NCT04137939
Title: Smart Health Care and Innovative Technology Service Model Plan : Development of Innovative Health Promotion System for Senior Adults
Brief Title: The Effect of IoT-based Smart Exercises System in the Senior Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B-BR-106-072
Record Dates: First submitted 2019-09-11; First posted 2019-10-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Elderly Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Ctrl group is instructed to maintain their original daily life
- Smart Exercise group (Experimental): SE group are instructed to perform one session of upper extremity ergometer and one session of lower extremity ergometer in a week, 30 minute per session, lasting for 12 weeks.
  Interventions: Device: smart exercise system

INTERVENTIONS:
Device: smart exercise system — The smart exercise system contains an upper extremity ergometer (UEE) and a lower extremity ergometer (LEE). The revolutions per minute (RPM) of the ergometer are instructed to maintain in 55-65. The resistance of UEE is set from level 1 at the first session, and adjusted by rating of perceived exertion (RPE) of each user after each end of the session. The resistance of LEE is set from level 2 at the first session, and adjusted by rating of perceived exertion (RPE) of each user after each end of the session.
  Arms: Smart Exercise group

SUMMARY:
Subjects are divided into two groups, (1) Control (Ctrl) and (2) Smart Exercise (SE) group. Ctrl group are instructed to maintain their daily life. SE participants are instructed to do exercise with smart exercise system twice per week for 12 weeks. The physical fitness tests and questionnaire of both group are performed before and after the 12-week exercise program.

DETAILED DESCRIPTION:
The smart exercise system contain an upper extremity cycle ergometer (UEE) and a lower extremity cycle ergometer (LEE). SE group are instructed to do once session of UEE and once session of LEE per week, 30 minute per session, lasting for 12 weeks. Before each exercise, the physiological parameter are measured to ensure safety. During exercise, heart rate of user and revolutions per minute (RPM) of the ergometer is detected per second. After each session of exercise, the rating of perceived exertion (RPE) of user is also inquired and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 50 years old
* No significant limb disability or joint deformation
* No history of cardiovascular disease
* Never lost balance due to dizziness in the past 12 months

Exclusion Criteria:

* limb disability or joint deformation
* history of cardiovascular disease
* lost balance due to dizziness in the past 12 months
* cognitive deficits

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
30 second chair stand test | baseline
  number of full stands that can be completed in 30 seconds with arms folded across chest.
30 second chair stand test | after 12-week intervention
  number of full stands that can be completed in 30 seconds with arms folded across chest.

SECONDARY OUTCOMES:
BMI | baseline
  Participant's weight in kilograms divided by the square of height in meters is recorded as Body Mass Index (BMI) .
BMI | after 12-week intervention
  Participant's weight in kilograms divided by the square of height in meters is recorded as Body Mass Index (BMI) .
SMI | baseline
  Skeletal muscle mass index (SMI), which is the sum of the muscle masses of the four limbs as appendicular skeletal mass (ASM) in kilograms divided by the square of height in meters, is detected by bioelectrical impedance analysis.
SMI | after 12-week intervention
  Skeletal muscle mass index (SMI), which is the sum of the muscle masses of the four limbs as appendicular skeletal mass (ASM) in kilograms divided by the square of height in meters, is detected by bioelectrical impedance analysis.
Back scratch | baseline
  Back scratch: with one hand reaching over the shoulder and one up the middle of the back, the distance(cm) between extended middle fingers is recorded.
Back scratch | after 12-week intervention
  Back scratch: with one hand reaching over the shoulder and one up the middle of the back, the distance(cm) between extended middle fingers is recorded.
Chair sit-&-reach test | baseline
  From a sitting position at front of chair, with leg extended and hands reaching toward toes, the distance(cm) between extended fingers and tip of toe is recorded.
Chair sit-&-reach test | after 12-week intervention
  From a sitting position at front of chair, with leg extended and hands reaching toward toes, the distance(cm) between extended fingers and tip of toe is recorded.
Six-minute walk test | baseline
  To walk as much as possible within six minutes and measure the total distance traveled.
Six-minute walk test | after 12-week intervention
  To walk as much as possible within six minutes and measure the total distance traveled.
2-minute step test | baseline
  2-minute step test is to complete steps in 2 minutes. Number of full steps completed in 2 minutes is recorded.
2-minute step test | after 12-week intervention
  2-minute step test is to complete steps in 2 minutes. Number of full steps completed in 2 minutes is recorded.
8-foot up-&-go test | baseline
  8-foot up-&-go test: number of seconds required to get up from a seated position, walk 8 feet, turn, and return to seated position.
8-foot up-&-go test | after 12-week intervention
  8-foot up-&-go test: number of seconds required to get up from a seated position, walk 8 feet, turn, and return to seated position.
Single leg balance with eyes open test | baseline
  Participant is instructed to stand by one leg with eye open, the number of seconds is recorded.
Single leg balance with eyes open test | after 12-week intervention
  Participant is instructed to stand by one leg with eye open, the number of seconds is recorded.
Hand grip strength test | baseline
  hand grip strength test is performed by HandGRIP Dynamometer to detect the grip strength
Hand grip strength test | after 12-week intervention
  hand grip strength test is performed by HandGRIP Dynamometer to detect the grip strength
SOF (Study of Osteoporotic Fractures) frailty index (Questionnaire for physical function and health status) | after 12-week intervention
  Risk factors for fractures and falls and has grown to look at various determinants of successful aging. Three questions about frailty and two questions about depression.
SOF (Study of Osteoporotic Fractures) frailty index (Questionnaire for physical function and health status) | baseline
  Risk factors for fractures and falls and has grown to look at various determinants of successful aging. Three questions about frailty and two questions about depression.
SARC-F | after 12-week intervention
  The SARC-F questionnaire is a Fast diagnostic test for SARCopenia. The questionnaire contains five items, which are Strength, Assistance in walking, Rise from a chair, Climb stairs, and Falls. The scores range from 0 to 10, with 0 to 2 points for each component. Score equal to or greater than 4 is predictive of sarcopenia and poor outcomes.
SARC-F | baseline
  The SARC-F questionnaire is a Fast diagnostic test for SARCopenia. The questionnaire contains five items, which are Strength, Assistance in walking, Rise from a chair, Climb stairs, and Falls. The scores range from 0 to 10, with 0 to 2 points for each component. Score equal to or greater than 4 is predictive of sarcopenia and poor outcomes.
EQ-5D (EuroQol- 5 Dimensions) | baseline
  EQ-5D is a standardized instrument with 5-item questionnaire for measuring generic health status. EQ-5D was first introduced in 1990 by the EuroQol Group. In which health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).
EQ-5D (EuroQol- 5 Dimensions) | after 12-week intervention
  EQ-5D is a standardized instrument with 5-item questionnaire for measuring generic health status. EQ-5D was first introduced in 1990 by the EuroQol Group. In which health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).
QUEST (Questionnaire for satisfaction) | after 12-week intervention
  The 8 items of the questionnaire included Dimensions, Weight, Ease in Adjusting, Safety and Security, Durability , Ease of Use, Comfortable, and Effectiveness. Each item employed a 5-point scale, with 1-point representing not satisfied at all, and 5-point representing very satisfied.Evaluation of Satisfaction with Assistive Technology

CONTACTS AND LOCATIONS:
Overall Officials: Li-Chieh Kuo, Ph. D., Study Director — National Cheng-Kung University Hospital
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan, Taiwan

REFERENCES:
- [Derived] Lin CC, Lin YS, Yeh CH, Huang CC, Kuo LC, Su FC. An Exergame-Integrated IoT-Based Ergometer System Delivers Personalized Training Programs for Older Adults and Enhances Physical Fitness: A Pilot Randomized Controlled Trial. Gerontology. 2023;69(6):768-782. doi: 10.1159/000526951. Epub 2023 Jan 6. PMID 36617413